CLINICAL TRIAL: NCT03159598
Title: Drain-Less Abdominally Based Breast Reconstruction Using a Novel Lysine-Derived Urethane Adhesive (TissueGlu, Cohera Medical)
Brief Title: Drain-Less Abdominally Based Breast Reconstruction Using Lysine-Derived Urethane Adhesive
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution, never submitted to IRB
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CASE5117
Record Dates: First submitted 2017-05-17; First posted 2017-05-18 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Breast Cancer
Keywords: A-BR; Abdominal-based breast reconstruction; Seroma
MeSH Terms: conditions — Breast Neoplasms; Seroma | interventions — Drainage; Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: This study has three parallel groups. One experimental and two control groups
Who Masked: Participant
Masking Description: The study is "semi-blind" in that patients will not be told which treatment they are receiving. If the patient is assigned to one of the drains groups, she will know post-operatively that she has drains, but she will not know if TissueGlu was utilized. The doctor will be aware of what treatment the patient is receiving, as he or she will administer the drug
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Tissue Glu with drains (Active Comparator): This is standard of care to use Tissue Glu in addition to a drain. Pre-operatively, as well as on post-operative patients will be asked to complete a questionnaire that addresses their pain, impact of drains on activities of daily living, social and physical activities. Patients will also be asked to provide information regarding who is caring for the drains, the impact of drains on the caregiver, the amount of anxiety the patient has related to drain removal and the amount of pain associated with drain removal
  Interventions: Device: Tissue Glu; Device: Drain; Other: Questionnaires
- Tissue Glu without drains (Experimental): This group utilizes Tissue Glu without the presence of a drain. Pre-operatively, as well as on post-operative patients will be asked to complete a questionnaire that addresses their pain, impact of drains on activities of daily living, social and physical activities. Patients will also be asked to provide information regarding who is caring for the drains, the impact of drains on the caregiver, the amount of anxiety the patient has related to drain removal and the amount of pain associated with drain removal
  Interventions: Device: Tissue Glu; Other: Questionnaires
- Drains (Active Comparator): This is standard of care to use traditional closed-suction drains. Pre-operatively, as well as on post-operative patients will be asked to complete a questionnaire that addresses their pain, impact of drains on activities of daily living, social and physical activities. Patients will also be asked to provide information regarding who is caring for the drains, the impact of drains on the caregiver, the amount of anxiety the patient has related to drain removal and the amount of pain associated with drain removal
  Interventions: Device: Drain; Other: Questionnaires

INTERVENTIONS:
Device: Tissue Glu — Once adequate hemostasis has been achieved during surgery and the abdominal fascia and flaps have been irrigated, Tissue Glu will be applied. Tissue Glu is applied at approximately one centimeter intervals while remaining one centimeter away from the umbilicus and inferior incisions.
  Other Names: TissuGlu; lysine-derived urethane adhesive
  Arms: Tissue Glu with drains; Tissue Glu without drains
Device: Drain — Drains will be placed during surgery to allow for the drainage of seroma which may develop after surgery
  Other Names: closed-suction drains
  Arms: Drains; Tissue Glu with drains
Other: Questionnaires — Questionnaires given to patients pre-and post surgery to determine pain, impact of breast reconstruction on activity, and impact of breast reconstruction on caregivers

SUMMARY:
Drains are routinely utilized in breast reconstruction when using abdominal tissue of the patient to remove fluid buildup while the body heals after surgery. However, drains are associated with patient discomfort, anxiety, decreased mobility, increased hospital stays and outpatient visits. Drains can also serve as a site of origin for infection as the system is not completely closed, and infectious organisms could theoretically use the drain as point of entry.

This proposed study investigates a potential novel mechanism to prevent the development of seromas (pockets of clear fluid which can develop after surgery) in patients who undergo breast reconstruction with their own abdominal tissue. By eliminating the required use of a drain, the study team expects patients to have less pain and use less pain medication, as well as more satisfaction with their overall surgical experience.

DETAILED DESCRIPTION:
Objectives:

1. Establish the safety of a lysine-derived urethane adhesive (TissuGlu, Cohera Medical) in patients undergoing autologous abdominal-based breast reconstruction. This will be assessed via analyzing complication profiles of patients post-operatively. The primary endpoints are rate of seroma development, need for seroma drainage and time to drain removal (if in drain group).
2. Determine if there is a difference in pain and other quality of life measures when comparing patients who do and do not have abdominal drains. This will be assessed via pain medicine utilization and by delivering a targeted survey pre-operatively, as well as at post-operative day three and four weeks.

Study Design:

Patients will be randomized to one of three arms: 1) Traditional closed-suction drains, 2) TissuGlu with closed-suction drains and 3) TissuGlu without closed-suction drains.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing Abdominally-Based Breast Reconstruction

  * Both unilateral or bilateral reconstruction is allowed
* Both delayed or immediate reconstruction is allowed

Exclusion Criteria:

* Diabetes
* BMI>30
* Active smokers.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Rate of seroma development | Up to 30 days after surgery
  Number of seromas which develop during the first 30 days after surgery.

SECONDARY OUTCOMES:
Difference in pain between patients with and without abdominal drains | Up to 4 weeks after surgery
  Patients will be given a questionnaire pre-operatively and the same questionnaire post-operatively. The change in these questionnaires will be compared between groups
Pain Medicine Utilization | Up to 4 weeks after surgery
  Use of pain medicine after surgery between groups, as indicated by chart review
Time to drain removal | Up to 4 weeks after surgery
  Time from surgery to the removal of the drain for any reason, in patients who were given a drain

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Moreira, MD, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center